CLINICAL TRIAL: NCT04127565
Title: Implementation Strategy From Research to Routine Care of a Comprehensive Prehospital Telemedicine System and Pre-post Analysis of Systemic Effects
Brief Title: Implementation Strategy and Systemic Effects of Routine Telemedical Care in Prehospital Emergency Medicine
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Dr. med. Sebastian Bergrath, Senior Physician, RWTH Aachen University
Other Study IDs: TNA2019-01
Record Dates: First submitted 2019-10-04; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Telemedicine Usage; Teleconsultation Usage; Emergency Medical Service Missions
Keywords: Telemedicine; Emergency Medical Service

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-implementation period: All emergency medical service missions (EMS) in the city of Aachen (Germany) from April 2013 to March 2014.
  Analysis of all ambulance calls and fraction of calls with support by an physician-staffed EMS unit, help of neighboring EMS units and helicopter emergency medical service units.
- Post-implementation period: All emergency medical service missions (EMS) in the city of Aachen (Germany) from April 2015 to March 2016.
  Analysis of all ambulance calls and fraction of calls with support by an physician-staffed EMS unit, help of neighboring EMS units and helicopter emergency medical service units.
  Additionally analysis of all ambulance calls with telemedical support.

SUMMARY:
In two research projects a comprehensive prehospital telemedicine system was developed and general feasibility as well as impact on guideline adherence were evaluated. These results allowed stepwise implementation into medical routine care.

All steps and milestones from the research idea to implementation were analyzed and evaluated descriptively in this study. Using a pre-post intervention analysis the systemic effects of the implementation on change in emergency medical resource utilization were analyzed.

DETAILED DESCRIPTION:
In two interdisciplinary research projects a comprehensive prehospital telemedicine system was developed and general feasibility as well as impact on guideline adherence were evaluated. Feasibility and general safety were demonstrated. These results allowed stepwise implementation into medical routine care during a one year phase. During implementation positive effects on guideline adherence were found. Despite positive results there are many barriers that prevent implementation of research projects into routine medical care. Therefore, the current study evaluated and interpreted all steps and milestones from the research idea to implementation and evaluated them descriptively. Using a pre-post intervention analysis the systemic effects of the implementation on change in emergency medical resource utilization were analyzed. Resource utilization of physician staffed emergency medical service units was compared between a pre-implementation period (12 months, April 2013 - March 2014) and a post-implementation period (12 months, April 2015 - March 2016). During the pre-implementation period only standard care was available.

Inclusion criteria: All emergency medical service (EMS) missions in both periods.

Data sources: Electronic health records of the EMS missions (data pseudonymity) and database of the regional EMS dispatch center.

ELIGIBILITY:
Inclusion Criteria:

All patients treated by emergency medical service during the pre- and post-implementation period.

Post-implementation period: Patients had to give verbal consent prior to teleconsultation.

Exclusion Criteria:

Pre-implementation period: none Post-implementation period: Patients who refused teleconsultation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pre-intervention period:
  Only standard care was provided. No patient data was obtained, only number of emergency calls and used resources were analyzed.
  Post-intervention period:
  Evaluation of conducted medical procedures in patients who received telemedical support (after given verbal consent). Number of emergency calls and used resources were compared to the pre-intervention period.
Sampling Method: Non-Probability Sample
Enrollment: 51649 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Change in usage of physician staffed EMS units | Comparison between 1 year pre-implementation and 1 year post-implementation period.
  Change in usage of physician staffed EMS units (ground based and helicopter based). Comparison between the pre- and post-implementation period.

SECONDARY OUTCOMES:
Usage of telemedical support in the post-implementation period | Through study completion in the post-implementation period (1 year)
  Number of ambulance calls using telemedical support
Provided medications during teleconsultation | Through study completion in the post-implementation period (1 year)
  Number of delegated medications including opioids in the post-implementation phase

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Rossaint, Prof. Dr., Study Director — University Hospital Aachen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergrath S, Muller M, Rossaint R, Beckers SK, Uschner D, Brokmann JC. Guideline adherence in acute coronary syndromes between telemedically supported paramedics and conventional on-scene physician care: A longitudinal pre-post intervention cohort study. Health Informatics J. 2019 Dec;25(4):1528-1537. doi: 10.1177/1460458218775157. Epub 2018 Jun 4. PMID 29865891
- [Background] Brokmann JC, Rossaint R, Muller M, Fitzner C, Villa L, Beckers SK, Bergrath S. Blood pressure management and guideline adherence in hypertensive emergencies and urgencies: A comparison between telemedically supported and conventional out-of-hospital care. J Clin Hypertens (Greenwich). 2017 Jul;19(7):704-712. doi: 10.1111/jch.13026. Epub 2017 May 30. PMID 28560799
- [Background] Lenssen N, Krockauer A, Beckers SK, Rossaint R, Hirsch F, Brokmann JC, Bergrath S. Quality of analgesia in physician-operated telemedical prehospital emergency care is comparable to physician-based prehospital care - a retrospective longitudinal study. Sci Rep. 2017 May 8;7(1):1536. doi: 10.1038/s41598-017-01437-5. PMID 28484212
- [Background] Brokmann JC, Conrad C, Rossaint R, Bergrath S, Beckers SK, Tamm M, Czaplik M, Hirsch F. Treatment of Acute Coronary Syndrome by Telemedically Supported Paramedics Compared With Physician-Based Treatment: A Prospective, Interventional, Multicenter Trial. J Med Internet Res. 2016 Dec 1;18(12):e314. doi: 10.2196/jmir.6358. PMID 27908843
- [Background] Felzen M, Brokmann JC, Beckers SK, Czaplik M, Hirsch F, Tamm M, Rossaint R, Bergrath S. Improved technical performance of a multifunctional prehospital telemedicine system between the research phase and the routine use phase - an observational study. J Telemed Telecare. 2017 Apr;23(3):402-409. doi: 10.1177/1357633X16644115. Epub 2016 Apr 13. PMID 27080747
- [Background] Brokmann JC, Rossaint R, Bergrath S, Valentin B, Beckers SK, Hirsch F, Jeschke S, Czaplik M. [Potential and effectiveness of a telemedical rescue assistance system. Prospective observational study on implementation in emergency medicine]. Anaesthesist. 2015 Jun;64(6):438-45. doi: 10.1007/s00101-015-0039-1. Epub 2015 Jun 3. German. PMID 26036316
- [Background] Rortgen D, Bergrath S, Rossaint R, Beckers SK, Fischermann H, Na IS, Peters D, Fitzner C, Skorning M. Comparison of physician staffed emergency teams with paramedic teams assisted by telemedicine--a randomized, controlled simulation study. Resuscitation. 2013 Jan;84(1):85-92. doi: 10.1016/j.resuscitation.2012.06.012. Epub 2012 Jun 30. PMID 22750663
- [Background] Skorning M, Bergrath S, Rortgen D, Beckers SK, Brokmann JC, Gillmann B, Herding J, Protogerakis M, Fitzner C, Rossaint R; Med-on-@ix-Working Group. Teleconsultation in pre-hospital emergency medical services: real-time telemedical support in a prospective controlled simulation study. Resuscitation. 2012 May;83(5):626-32. doi: 10.1016/j.resuscitation.2011.10.029. Epub 2011 Nov 22. PMID 22115932
- [Background] Bergrath S, Rortgen D, Rossaint R, Beckers SK, Fischermann H, Brokmann JCh, Czaplik M, Felzen M, Schneiders MT, Skorning M. Technical and organisational feasibility of a multifunctional telemedicine system in an emergency medical service - an observational study. J Telemed Telecare. 2011;17(7):371-7. doi: 10.1258/jtt.2011.110203. Epub 2011 Sep 20. PMID 21933897
- [Derived] Bergrath S, Brokmann JC, Beckers S, Felzen M, Czaplik M, Rossaint R. Implementation of a full-scale prehospital telemedicine system: evaluation of the process and systemic effects in a pre-post intervention study. BMJ Open. 2021 Mar 24;11(3):e041942. doi: 10.1136/bmjopen-2020-041942. PMID 33762230